CLINICAL TRIAL: NCT00409552
Title: Phase 1 and 2 Study of Human Factors Analysis in VR for Burn Treatment
Brief Title: Human Factors Analysis in VR for Burn Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N44DA-5-7744
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2009-09

CONDITIONS: Pain; Chronic Pain
MeSH Terms: conditions — Pain; Chronic Pain

ARMS (5):
- 1 (Experimental): Virtual Reality with head display
  Interventions: Behavioral: Virtual Reality based distraction
- 2 (Active Comparator): Virtual Reality with flat projection display
  Interventions: Behavioral: VR with flat projection display
- 3 (Active Comparator): non-interactive video with head display
  Interventions: Behavioral: non-interactive video with head display
- 4 (Active Comparator): non-interactive video with flat projection display
  Interventions: Behavioral: non-interactive video with with flat projection display
- 5 (No Intervention): No distraction

INTERVENTIONS:
Behavioral: Virtual Reality based distraction — Participants will undergo virtual reality based distraction using the head display while they go through the pain process.
  Arms: 1
Behavioral: VR with flat projection display — VR with flat projection display
  Arms: 2
Behavioral: non-interactive video with head display — non-interactive video with head display
  Arms: 3
Behavioral: non-interactive video with with flat projection display — non-interactive video with with flat projection display
  Arms: 4

SUMMARY:
A number of studies have shown that virtual reality (VR) can be used to distract patients from pain and anxiety during painful medical procedures for which medication provides inadequate relief. An inexpensive, commercially available VE could have significant impact in reducing perceived pain involved in a variety of medical procedures. The Virtual Reality Medical Center (VRMC) developed an engaging virtual world that proved to be effective in reducing reported pain ratings of participants experiencing several different forms of painful stimuli. The virtual world called Icy Cool World was found to successfully distract patients from painful stimuli and reduce patients' perceived levels of pain. Phase II looks to expand on these findings and examine the effectiveness as a pain distraction technique for a variety of acute and chronic pain etiologies. The main objective of the clinical investigation will be to expand on the findings from earlier studies and obtain a more comprehensive analysis regarding the clinical versatility of VR pain distraction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65, male or female, any ethnicity as long as candidates can understand and read English adequately.

Exclusion Criteria:

* We will exclude participants who meet DSM-IV-TR criteria for alcohol or other substance abuse in the past year, or are currently using any recreational drugs, or taking more than 20 alcoholic drinks a week. In addition, the Beck Depression Inventory II (BDI-II) score must be less than 16, with no suicidal ideation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pain rating reduction | Following each trial

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Wiederhold, MD, PhD, FACP, Principal Investigator — VRMC